CLINICAL TRIAL: NCT07197268
Title: An Open-Label Single Center, Single Participant Study of an Experimental Antisense Oligonucleotide Treatment for Bainbridge-Ropers Syndrome Due to ASXL3 Gene Variant
Brief Title: Personalized Antisense Oligonucleotide Therapy for A Single Participant With ASXL3 Gene Mutation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-0542
Record Dates: First submitted 2025-07-24; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-07

CONDITIONS: Bainbridge-Ropers Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-ASXL3-001

INTERVENTIONS:
Drug: nL-ASXL3-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with Bainbridge-Ropers Syndrome (BRPS) due to a pathogenic, de novo nonsense variant in ASXL3

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with BRPS due to a pathogenic, de novo nonsense variant in ASXL3

ELIGIBILITY:
Inclusion Criteria:

* Informed consent/assent provided by the participant (when appropriate), and/or participant's parent(s) or legally authorized representative(s)
* Ability to travel to the study site and adhere to study-related follow-up examinations and/or procedures and provide access to participant's medical records
* Genetically confirmed ASXL3 genetic variant

Exclusion Criteria:

* Participant has any condition that, in the opinion of the Site Investigator, would ultimately prevent the completion of stud procedures

Ages: 4 Years to 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2025-05-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to 24 months
  Incidence and severity of treatment-emergent adverse events (AEs) from baseline to 12- and 24-months post nL-ASXL3-001 administration
Safety and Tolerability | Baseline to 24 months
  Changes from baseline to 12- and 24-months post nL-ASXL3-001 administration in physical examination (changes in appearance, skin, neck, ears, nose, throat, heart/lungs, abdomen, lymph nodes, and extremities compared to baseline)
Incidence of Treatment Emergent Abnormalities in Neurological Exam [Safety and Tolerability] | Baseline to 24 months
  Changes from baseline to 12- and 24-months post nL-ASXL3-001 administration in neurological examination (changes in mental status, gait, cerebellar, cranial nerve, motor, reflex, and sensations compared to baseline)
Incidence of Treatment-Emergent Abnormalities in Safety Labs (CSF, chemistry, hematology, coagulation, urinalysis) [Safety and Tolerability] | Baseline to 24 months
  Emergent abnormalities in laboratory analyses (results outside of normal range for CSF, chemistry, hematology, coagulation, and urinalysis)
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-ASLX3-001 administration as measured by the Vineland Adaptive Behavior Scales - Third Edition (Vineland-3) score.
Motor Skills | Baseline to 24 months
  Change in gross motor function from baseline to 12- and 24-months post nL-ASXL-001 administration as measured by the Gross Motor Function Measure (GMFM 88/66)

SECONDARY OUTCOMES:
Feeding Tolerance and Growth | Baseline to 24 months
  Change in feeding tolerance and growth from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by body mass index (BMI).
Feeding tolerance and growth | Baseline to 24 months
  Change in feeding tolerance and growth from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by % oral feeding vs G tube reported by parent feeding diary
Feeding tolerance and growth | Baseline to 24 months
  Change in feeding tolerance and growth from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by Functional Oral Intake Score (FOIS)
Feeding Tolerance and Growth | Baseline to 24 months
  Change in feeding tolerance and growth from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by Bristol Stool Scale
Cognition, Communication, and Behavior | Baseline to 24 months
  Change in communication from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by Vineland Adaptive Behavior Scales - Third Edition (Vineland-3): growth scale values (GSVs) for Expressive Language and Receptive Language subdomains
Cognition, Communication, and Behavior | Baseline to 24 months
  Change in cognition, communication, and behavior from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by Bayley Scales of Infant and Toddler Development 4th Edition (BSID-4): Expressive and Receptive Language Domains and Receptive Language Domains and Cognition Domain
Cognition, Communication, and Behavior | Baseline to 24 months
  Change in cognition, communication, and behavior from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by Observer-Related Communication Ability (ORCA) overall T score
Cognition, Communication, and Behavior | Baseline to 24 months
  Change in cognition, communication, and behavior from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by Aberrant Behavior Checklist (ABC)
Cognition, Communication, and Behavior | Baseline to 24 months
  Change in cognition, communication, and behavior from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by Repetitive Behavior Scale
Quality of Life | Baseline to 24 months
  Change in quality of life from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by the Quality-of-Life Inventory - Disability (QI-Disability)

OTHER OUTCOMES:
Swallow Function | Baseline to 24 months
  Change in swallowing function from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by video fluoroscopic swallow study (VFSS)
Swallow Function | Baseline to 24 months
  Change in swallowing function from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by modified barium swallow study (MBSS)
Vision | Baseline to 24 months
  Change in vision from baseline to 12- and 24-months post nL-ASXL3-001 administration as measured by cortical vision impairment assessment
Sleep | Baseline to 24 months
  Change in Sleep from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by parent-reported sleep diary
Sleep | Baseline to 24 months
  Change in Sleep from baseline to 6-, 12-, 18-, and 24-months post nL-ASXL3-001 administration as measured by Sleep Disturbances Scale for Children (SDSC)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina Chapel Hill, Chapel Hill, North Carolina, United States